CLINICAL TRIAL: NCT06379230
Title: A Retrospective Study on Epidemiological Characteristics of Chinese NF1 Patients in Real World (PROMISE)
Status: Recruiting | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: SH9H-2023-T378-1
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Neurofibromatosis 1; Plexiform Neurofibroma
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This study is purely descriptive study. — This study is purely descriptive study.

SUMMARY:
Background/Rationale: Neurofibromatosis type 1 (NF1) affects about 1 in every 3000 people worldwide. Globally, 30~50% NF1 patients will develop plexiform neurofibromas (PNs), which grow rapidly in early childhood and can cause disfigurement, motor dysfunction, pain, airway dysfunction, visual impairment and bladder and bowel dysfunction. This systemic disease imposes a heavy psychosomatic and financial burden on patients and their caregivers. In NF1 patients, the lifetime risk of MPNST developed from PN is 8% to 13%. The mean age for NF1-associated death was approximately 20 years lower than that for the general population. Limited epidemiological and clinical data of Chinese NF1 patients is available to date. And the treatment pattern of Chinese NF1-PN patients is also unknown.

Objectives and Hypotheses: It is a descriptive study without formal hypothesis. The primary objective of this study is determining the percentage of NF1 patients who develop PN. The secondary objectives of this study include describing the clinical characteristics, tumor progression and treatment pattern of NF1-PN. The exploratory objective is exploring the epidemiological characteristics of other NF1 manifestations.

Methods:

Study design: The study is a retrospective multi-center chart review study. Data Source(s): All the data will be collected by CRF from inpatient and outpatient electronic medical records in every study site from January 1, 2019 to December 31, 2022.

Study Population: Patients who attended the study sites between January 1, 2019 - December 31, 2022 and were diagnosed with NF1 were included in this study. Statistical Analysis: This study is purely descriptive without any formal hypotheses.

Missing data for baseline characteristics will be assessed and addressed as a categorical variable with a level for missingness. All reported measures will be summarized in the study tables. Point estimates and their 95% CIs will be presented in the final analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who attended the study sites between January 1, 2019, and December 31, 2022.
2. Patients who were diagnosed with NF1(recorded with the text of type I neurofibromatosis) based on National Institutes of Health (NIH) NF1 consensus.

Exclusion Criteria:

1. Patients combined with other malignant tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be included in this study if they: 1) attended the study sites between January 1, 2019 and December 31, 2022; 2) were diagnosed with NF1 based on NIH NF1 consensus (Version 1987 or Version 2021); and 3) were not diagnosed with other malignant tumors from 2019.1.1 to 2022.12.31. As this study was a chart review, there was no systematic follow-up. Follow-up was based on individual patient needs, was not dictated by the study, and varied from person to person in a manner reflective of real clinical practice. Thus, patients were followed up until end of data availability, death, or loss of follow up, whichever comes first.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Determine the percentage of NF1 patients developed PN at the baseline. | 2022.12.31
  The clinical diagnosis of PN mainly depends on the clinical manifestations and imaging of NF1 patients. Superficial PN has a clear clinical manifestation. It refers to a proliferation of cells in the nerve sheath which involves multiple nerve fascicles, forming a large pendulous mass with skin pigmentation on the surface. PN in vivo often has no significant clinical features and requires imaging examination, like MRI. Patients diagnosed with PN are recorded with the text of plexiform neurofibromas in the chart.
  The percentage of patients diagnosed with PN with imaging and the percentage of patients diagnosed with PN without imaging will be calculated.

SECONDARY OUTCOMES:
Clinical characteristics of NF1-PN: | 2022.12.31
  Describe the percentage of symptomatic NF1-PN at the baseline.
Tumor progression of NF1-PN | 2022.12.31
  Describe the 1-year/2-year/3-year progression-free survival (PFS) rate of NF1- PN.
Treatment pattern of NF1-PN: | 2022.12.31
  Describe the percentage of NF1-PN patients underwent surgeries after index date.

OTHER OUTCOMES:
The exploratory endpoints: | 2022.12.31
  Epidemiological characteristics of other NF1 manifestations:
  Describe the percentage of NF1 patients with cNF at the baseline.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No